CLINICAL TRIAL: NCT04576689
Title: RIPPLE-1: Evaluation of Safety and Efficacy of the IBE-814 Intravitreal Implant in Patients with Diabetic Macular Oedema and Macular Oedema Due to Retinal Vein Occlusion
Brief Title: Safety and Efficacy of IBE-814 Intravitreal (IVT) Implant - a Sustained, Low Dose Dexamethasone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ripple Therapeutics Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Organization: Ripple Therapeutics Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBE-814-IVT-1
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Macular Oedema; Retinal Vein Occlusion with Macular Oedema
MeSH Terms: interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose (Experimental): One (1) IBE-814 IVT Implant (70 μg Dexamethasone) Route of administration: intravitreal injections
  Interventions: Drug: IBE-814 70ug
- High dose (Experimental): Two (2) IBE-814 IVT Implant (140 μg Dexamethasone) Route of administration: intravitreal injections
  Interventions: Drug: IBE-814 140ug

INTERVENTIONS:
Drug: IBE-814 70ug — At least 10 and up to 33 participants will receive one (1) IBE-814. Route of administration: intravitreal injection.
  Other Names: Low dose
  Arms: Low dose
Drug: IBE-814 140ug — Up to 27 participants will receive two (2) IBE-814. Route of administration: intravitreal injection.
  Other Names: High dose
  Arms: High dose

SUMMARY:
This trial is a phase II, multi-center, single-masked (assessors) dose-ranging study designed to evaluate the comparative safety and preliminary efficacy of two dosage regimens of the IBE-814 IVT Dexamethasone Implant in patients with DMO and RVO.

DETAILED DESCRIPTION:
The study will enroll up to 60 patients (up to 60 eyes) with DMO or RVO across two treatment groups (Low Dose and High Dose). Patients will be identified and recruited through the clinic population of ophthalmology centers in Australia, New Zealand, Hong Kong, and Canada specializing in the diagnosis and treatment of retinal diseases. All patients will be followed for a planned evaluation period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years at the time of informed consent
* Able and willing to provide informed consent
* A diagnosis of CRVO defined as: The study eye has retinal hemorrhage or other biomicroscopic evidence of RVO (e.g. telangiectatic capillary bed) and a dilated venous system (or previously dilated venous system) in all four quadrants AND Retinal thickening due to RVO involving the center of the macula of the study eye OR
* A diagnosis of BRVO defined as: The study eye has retinal hemorrhage or other biomicroscopic evidence of RVO (e.g. telangiectatic capillary bed) and a dilated venous system (or previously dilated venous system) in one quadrant or less of retina drained by the affected vein AND Retinal thickening due to RVO involving the center of the macula of the study eye OR
* A diagnosis of HRVO defined as: The study eye has retinal hemorrhage or other biomicroscopic evidence of RVO (e.g. telangiectatic capillary bed) and a dilated venous system (or previously dilated venous system) in two adjacent quadrants of retina drained by the affected vein AND Retinal thickening due to RVO involving the center of the macula of the study eye OR
* A diagnosis of diabetes mellitus (Type 1 or type 2) defined as one or more of the following: a) Current regular use of insulin for the treatment of diabetes, b) Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes, c) Documented diabetes by ADA and/or WHO (World Health Organization) criteria, AND Retinal thickening due to DMO involving the center of the macula of the study eye.
* The study eye meets all of the following criteria:

  1. Visual acuity letter score in study eye ≤73 and ≥24 (approximate Snellen equivalent 20/40 to 20/320).
  2. Patient has CST of at least 300 μm (by Cirrus/Spectralis) if measured by Cirrus OCT or 325 μm if measured by Spectralis OCT, with presence of intraretinal and/or subretinal fluid at Screening visit and within 14 days of the baseline treatment visit.
  3. Media clarity, pupillary dilation, and individual cooperation sufficient for adequate OCTs.
  4. Study eye has not received any prior intravitreal injections of anti-VEGF or steroids (i.e., treatment naïve).

OR

* Study eye has documented OCT evidence of an intravitreal anti-VEGF or steroid response with respect to macular oedema in the past 9 months. The response is defined as either a reduction of 30% or more of excess macular thickness or a reduction of 50 μm or greater. Excess macular thickness is defined as the amount of CST greater than 250 μm (by Cirrus/Spectralis).
* Must agree to use highly effective, medically accepted double-barrier contraception (both WOCBP and male partners of WOCBP) from Screening and for 12 months after last dose of study drug as specified below in this criterion.

Highly effective double-barrier contraception is defined as use of a condom AND one of the following:

1. Birth control pills (The Pill)
2. Depot or injectable birth control
3. IUD (Intrauterine Device)
4. Birth Control Patch
5. NuvaRing
6. Implantable contraception (e.g., Implanon)
7. Documented evidence of surgical sterilization at least 6 months prior to Screening, i.e., tubal ligation or hysterectomy for women or vasectomy for men

Rhythm methods are not considered as highly effective methods of birth control. Male subjects must refrain from sperm donation from start of study and for 12 months after the last dose of study drug. Subjects who are in same-sex relationships are not required to use contraception. Contraception does not apply to postmenopausal females (i.e. FSH ≥30 mIU/mL and ≥12 months since last menstruation).

Exclusion Criteria:

* Known allergy or hypersensitivity to corticosteroids or any component of the study treatments (including povidone iodine prep) including any prior fluorescein allergic reaction graded above mild or that was not adequately resolved with oral or topical medication.
* Active or suspected ocular or periocular infection
* History of steroid-induced IOP elevation to ≥30 mmHg that required IOP-lowering treatment
* Systemic steroid treatment within 4 months prior to enrollment or anticipated use during the study
* Initiation of intensive insulin treatment (a pump or multiple daily injections) within 4 months prior to randomization or plans to do so in the next 4 months
* Systolic blood pressure > 180mmHg or diastolic blood pressure > 110 mmHg
* Screening glycated hemoglobin (HbA1c) blood test >12.0%
* History of chronic renal failure requiring dialysis or kidney transplant
* Participation in an investigational trial within 30 days of enrolment that involved treatment with any drug that has not received regulatory approval for the indication being studied or participation in an investigational trial during this trial that may significantly impact safety and/or efficacy evaluations.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 3 months prior to enrolment
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 24 months.
* A condition that, in the opinion of the Investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control)
* Individual is expecting to move from the area of the study center to an area not covered by another center during the 18 months following randomization

For the study eye only:

* Posterior capsule of the lens is absent, torn, ulcerated or perforated due to any cause, except if due to YAG capsulotomy.
* Aphakia or anterior chamber IOL
* For patients with RVO in the study eye, presence of diabetic retinopathy in either eye
* Macular oedema is considered to be due to a cause other than DMO or RVO
* Macula is non-perfused on Screening fluorescein angiography.
* An ocular condition is present (e.g., foveal atrophy, pigment abnormalities, dense sub-foveal hard exudates, visually significant cataract, non-retinal condition, etc.), such that visual acuity loss would not improve from resolution of macular oedema.
* An ocular condition is present (other than DMO or RVO) that, in the opinion of the Investigator, might affect macular oedema or alter visual acuity during the study period (e.g., uveitis or other inflammatory eye disease, neovascular glaucoma, etc.), or it is expected that the patient will require a procedure within 24-weeks post-enrolment that may affect macular oedema or alter visual acuity (e.g., retinal photocoagulation treatment). After 24 weeks of enrolment, procedures may be performed after notifying the Sponsor and Medical Monitor.
* Presence of an epiretinal membrane or vitreo-retinal interface changes in the study eye which, in the opinion of the Investigator, is the primary cause of macular oedema, or is severe enough to prevent improvement in visual acuity despite reduction in macular oedema
* Substantial posterior capsule opacity that, in the opinion of the Investigator, is likely to be decreasing visual acuity by three lines or more (i.e., opacity would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* IOP greater than 21 mmHg while treated with more than one topical medical therapy.
* A documented diagnosis of glaucoma or IOP>21 mmHg and presence of glaucomatous optic nerve head observed by fundus examination.
* History of intraocular corticosteroid injection or implant within 6 months prior to study treatment.
* History of greater than one (1) OZURDEX® dexamethasone implant for phakic patients only. There is no limit for pseudophakic patients.
* History of IVT anti-VEGF injections within 6 weeks prior to study treatment.
* Any history of treatment with Retisert, Iluvien or Yutiq insert for phakic patients, or any treatment with Retisert, Iluvien or Yutiq in the previous 36 months for pseudophakic patients.
* History of macular laser photocoagulation within 4 months prior to study treatment.
* Any history of vitrectomy.
* History of cataract surgery within 3 months of enrolment or predicted within 6 months post-enrolment.
* History of YAG laser posterior capsulotomy within 3 months of enrolment or predicted within 6 months post-enrolment, or a prior YAG capsulotomy that does not sufficiently cover the borders of the IOL optic.
* Anterior capsule requires treatment for concurrent phimosis.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | Measurements from baseline to 6 months (24 weeks)
  Mean change in LogMAR best corrected visual acuity in the study eye
Central Subfield Thickness | Measurements from baseline to 6 months (24 weeks)
  Mean change in central subfield thickness on optical coherence tomography
Ocular and Non-Ocular Treatment Emergent Adverse Events | Baseline through 18 months
  Number of ocular and non-ocular treatment emergent adverse events, summarized at the patient level by system organ class and preferred term
Study Drug-Related Ocular Adverse Events | Baseline through 18 months
  The number of study drug-related ocular adverse events, summarized separately for study and fellow eyes, by system organ class and preferred term
Drug-Related Adverse Events | Baseline through 18 months
  Drug-related adverse events including: a) any new rise in intraocular pressure >27 mmHg in the study eye, at any visit; b) requirement for additional neuroprotective or IOP-lowering therapy, at any visit; c) requirement for surgery to reduce IOP, at any visit; d) any new diagnosis of cataract or significant lens opacification at any visit, significant worsening of cataract in the study eye during the study.
Post-Injection Complications | Baseline through 18 months
  Post-injection complications including worsening visual acuity, change in vision, worsening macular oedema, vitreous hemorrhage, retinal tear or detachments, inflammation, IOP alterations
Adverse Events | Baseline through 18 months
  Frequency and severity of adverse events throughout the primary outcome assessment period

CONTACTS AND LOCATIONS:
Overall Officials: Jagjit Gilhotra, Principal Investigator — Royal Adelaide Hospital
Locations (21):
- Australia (15):
  - Retina and Eye Consultants, Hurstville, New South Wales
  - Eye Doctors Mona Vale, Mona Vale, New South Wales
  - Marsden Eye Specialist, Parramatta, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic, Sydney, New South Wales
  - Newcastle Eye Hospital, Waratah, New South Wales
  - Queensland Eye Institute, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Armadale Eye Clinic, Malvern, Victoria
  - Eye Surgery Associates, Malvern, Victoria
  - Lions Eye Institute, Nedlands, Western Australia
- Canada (3):
  - Upton Eye Specialists, Brampton
  - Retina Centre Of Ottawa, Ottawa
  - Uptown Eye Specialists, Vaughan
- Hong Kong (2):
  - Grantham Hospital, Aberdeen
  - Prince of Wales Hospital the Chinese University of Hong Kong, Hong Kong
- Southern Eye Specialists, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romano F, Lamanna F, Gabrielle PH, Teo KYC, Battaglia Parodi M, Iacono P, Fraser-Bell S, Cornish EE, Nassisi M, Viola F, Agarwal A, Samanta A, Chhablani J, Staurenghi G, Invernizzi A. Update on Retinal Vein Occlusion. Asia Pac J Ophthalmol (Phila). 2023 Mar-Apr 01;12(2):196-210. doi: 10.1097/APO.0000000000000598. Epub 2023 Feb 14. PMID 36912792